CLINICAL TRIAL: NCT05812261
Title: Lesion Characteristics After Pulsed-Field Ablation in Patients With Atrial Fibrillation and a Left Common Ostium
Acronym: PFALCO Remap
Status: Completed | Type: Observational
Sponsor: Onze Lieve Vrouwe Gasthuis (Other)
Collaborators: OLVG (Network)
Responsible Party: Principal Investigator, Daniel Mol, Principal Investigator, Onze Lieve Vrouwe Gasthuis
Other Study IDs: WO.23.038
Record Dates: First submitted 2023-04-02; First posted 2023-04-13 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Atrial Fibrillation; Pulmonary Vein Isolation; Ablation Therapy
Keywords: Atrial fibrillation; Pulmonary vein isolation; Left common ostium; Pulsed-field ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Creating an electro-anatomical map — After the routine pulsed-field ablation procedure, the operator will create an electro-anatomical map using the ablation catheter and a 3D mapping system.

SUMMARY:
This study aims to investigate the lesion characteristics after pulmonary vein isolation using pulsed-field ablation in patients with atrial fibrillation and a common of the left pulmonary veins.

The main question it aims to answer is: In which percentage of the patients will pulsed field ablation result in successful isolation of the left common ostium?

Nineteen patients will be prospectively included in OLVG. All patients will be treated with pulsed-field ablation (routine care). After the ablation procedure, an electro-anatomical map will be created using the ablation catheter and a mapping system. This map will display the left atrium and the lesion in detail.

After the procedure, three experienced operators are asked to draw a line around the LCO in the anatomical map where they would have ablated if conventional radiofrequency ablation was used. The distance between the drawn line and the ablation lesion will be measured at three predefined points. The lesion is considered successful if the mean distance is within ±10mm at all measurement points.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common arrhythmia affecting millions worldwide with increasing prevalence. Patients with AF tend to have more comorbidity and an increased stroke and mortality risk. Pulmonary vein isolation (PVI) has become the cornerstone in the invasive treatment of atrial fibrillation (AF). It has been shown that PVI is more effective in maintaining sinus rhythm and improving quality of life compared to antiarrhythmic drugs. Although PVI results in a 98% burden reduction, an AF recurrence is observed in about half of the patients. AF type, comorbidity, and anatomical pulmonary vein variants affect arrhythmia-free survival.

Eighteen per cent of the patients undergoing PVI have a left common ostium (LCO) of the pulmonary veins.(16) A large ostium characterises an LCO, and single-shot devices tend to have worse arrhythmia-free survival than conventional radiofrequency (C-RF) ablation. A proper pulmonary vein occlusion is crucial during cryoballoon ablation. A large ostium can form a distal lesion with the possibility of pulmonary vein potentials proximal to the lesion resulting in AF recurrence. Wide antrum isolation has been shown to improve outcomes, and a distally located lesion can explain the higher AF recurrence rate.(18)

Farapulse (Boston Scientific, MA, US) pulsed-field ablation (PFA) was recently introduced. PFA uses short pulses of high voltages to achieve electroporation and irreversible cell membrane damage.(19) This technique is tissue-specific and limits collateral damage. While PV reconnection has been observed in 47% of patients who underwent cryoballoon or radiofrequency ablation, PFA ablation creates durable lesions in 86% of patients.(19, 20)

Tissue contact is less critical during PFA than conventional RF or cryoballoon ablation. Therefore one could hypothesise that, in patients with an LCO, PFA can be performed at the actual pulmonary vein ostium and that the lesion location is comparable to conventional RF ablation. Reddy et al. included patients with an LCO and presented an electro-anatomical map showing antral isolation. However, it is still being determined how many patients with an LCO were included, and a comprehensive description of the lesion still needs to be provided. Because no studies investigated the lesion characteristic in patients with AF and an LCO after PFA ablation, this study is designed to examine the lesion location in detail with an electro-anatomical map.

This single-centre study will be conducted prospectively in OLVG, Amsterdam, the Netherlands. Patients are eligible for this study if they are admitted for AF ablation because of symptomatic and drug-resistant/intolerant AF and have an LCO (identified by computer tomography (CT) or magnetic resonance imaging (MRI)). All inclusion and exclusion criteria are described in the paragraph ELIGIBILITY.

The operator will map the left atrial voltage in nineteen patients using the Ensite Precision (Abbott inc. IL, US) and the Farawave ablation catheter. First, all patients will be treated with pulsed-field ablation (routine care). Then, when all pulmonary veins are considered isolated, an electro-atomical map of the left atrium will be created.

After the procedure, three experienced operators are asked to draw a line in the anatomical map where they would have performed ablation if C-RF had been used - again, blinded for voltage. Next, the investigators will measure the distance between the line the operators drew and the ablation lesion at three points. The lesion is considered within range if the mean difference is ±10mm at all measurement points.

All study outcomes are specified in the paragraph OUTCOME MEASURES.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years of age on the day of enrolment of either sex
* Willing to the sign informed consent
* Left atrial volume index measured < 60 ml/m2 within last 12 months
* Documented atrial fibrillation
* Admitted and accepted for PVI
* A left common ostium of the pulmonary veins identified by CT or MRI
* Accepted to receive general anaesthesia

Exclusion Criteria:

* Patients aged < 18
* Body mass index > 35kg/m2
* Left atrial volume index ≥ 60 ml/m2 within 12 months on MRI or cardiac echo
* New York Heart Association heart failure class III or IV
* Myocardial infarction within three months before the procedure
* Unstable angina pectoris
* Percutaneous coronary interventions within three months before the procedure
* Sudden cardiac death event within three months before the procedure
* A life expectancy of less than one year
* Presence of an atrial tachycardia other than cavotricuspid isthmus-dependent atrial flutter
* History of blood clotting or bleeding abnormalities
* History of a thromboembolic event within six months before the procedure
* A contraindication to anticoagulant
* Clinical significant infection
* Unstable clinical significant medical condition
* Previous left atrium ablation, except successful accessory pathway ablation
* Presence of a left appendage closure device
* Presence of an atrial septum occluder
* Presence of a prosthetic heart valve
* Occlusion of the inferior venous tract
* Enrolment in another study that would interfere with this study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation and a common ostium of the left pulmonary veins admitted and accepted for pulsed-field ablation at OLVG, Amsterdam, will be enrolled if eligible.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2023-07-19 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Successful left common ostium isolation after pulsed-field ablation in patients with atrial fibrillation | Within one week after the procedure
  The distance between the lesion and the line drawn in the electro-anatomical map by three operators will be measured at three predefined points. The lesion is considered successful if the mean distance is within 10mm at all points.

SECONDARY OUTCOMES:
Successful isolation at each measuring point | Within one week after the procedure
  The mean distance between the lesion and line in the electro-anatomical map for each measuring point. (Superior roof, mid posterior, and inferior)
Distance between the left and right lesion | Within one week after the procedure
  Distance between the left and right lesion measured at the superior roof, mid posterior, and inferior
Correlation between posterior wall conduction speed and the left and right lesion distance | Within one week after the procedure
  Conduction speed at the posterior wall will be measured with an activation map. All the activation data will be collected simultaneously with the electro-anatomical map.
Safety outcomes within the hospital stay | 24 hours
  The occurrence of procedural-related complications, including:
  * Vascular complication (defined as a major or minor vascular complication from the Valve Academic Research Consortium-2)
  * Bleeding complication (defined as Bleeding Academic Research Consortium type 2 or higher)
  * Tamponade, for which an intervention is required
  * Transient phrenic nerve palsy (lasting < 24 hours)
  * Persistent phrenic nerve palsy (lasting ≥ 24 hours)
  * Thromboembolic event
  * Admission for more than 24 hours post-procedure and the reason for prolonged admission.
Number of patients with successful same-day discharge | 24 hours
  The number of patients who were successfully discharged and data on hospital prolongation will be collected.
Interoperator variability of the line drawn in the anatomical map | Within one week after the procedure
  The investigators will investigate the variation of the line drawn by three operators
True pulmonary vein isolation demonstrated with the Boston Farawave and Ensite Precision | During the procedure
  Here the investigators will investigate whether all pulmonary veins are isolation based on the information from the electro-anatomical map.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Mol, PhD, Principal Investigator — OLVG
Locations (1):
- OLVG, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data can be shared on reasonable request.

REFERENCES:
- [Background] Krijthe BP, Kunst A, Benjamin EJ, Lip GY, Franco OH, Hofman A, Witteman JC, Stricker BH, Heeringa J. Projections on the number of individuals with atrial fibrillation in the European Union, from 2000 to 2060. Eur Heart J. 2013 Sep;34(35):2746-51. doi: 10.1093/eurheartj/eht280. Epub 2013 Jul 30. PMID 23900699
- [Background] Odutayo A, Wong CX, Hsiao AJ, Hopewell S, Altman DG, Emdin CA. Atrial fibrillation and risks of cardiovascular disease, renal disease, and death: systematic review and meta-analysis. BMJ. 2016 Sep 6;354:i4482. doi: 10.1136/bmj.i4482. PMID 27599725
- [Background] Packer DL, Mark DB, Robb RA, Monahan KH, Bahnson TD, Poole JE, Noseworthy PA, Rosenberg YD, Jeffries N, Mitchell LB, Flaker GC, Pokushalov E, Romanov A, Bunch TJ, Noelker G, Ardashev A, Revishvili A, Wilber DJ, Cappato R, Kuck KH, Hindricks G, Davies DW, Kowey PR, Naccarelli GV, Reiffel JA, Piccini JP, Silverstein AP, Al-Khalidi HR, Lee KL; CABANA Investigators. Effect of Catheter Ablation vs Antiarrhythmic Drug Therapy on Mortality, Stroke, Bleeding, and Cardiac Arrest Among Patients With Atrial Fibrillation: The CABANA Randomized Clinical Trial. JAMA. 2019 Apr 2;321(13):1261-1274. doi: 10.1001/jama.2019.0693. PMID 30874766
- [Background] Mark DB, Anstrom KJ, Sheng S, Piccini JP, Baloch KN, Monahan KH, Daniels MR, Bahnson TD, Poole JE, Rosenberg Y, Lee KL, Packer DL; CABANA Investigators. Effect of Catheter Ablation vs Medical Therapy on Quality of Life Among Patients With Atrial Fibrillation: The CABANA Randomized Clinical Trial. JAMA. 2019 Apr 2;321(13):1275-1285. doi: 10.1001/jama.2019.0692. PMID 30874716
- [Background] Andrade JG, Champagne J, Dubuc M, Deyell MW, Verma A, Macle L, Leong-Sit P, Novak P, Badra-Verdu M, Sapp J, Mangat I, Khoo C, Steinberg C, Bennett MT, Tang ASL, Khairy P; CIRCA-DOSE Study Investigators. Cryoballoon or Radiofrequency Ablation for Atrial Fibrillation Assessed by Continuous Monitoring: A Randomized Clinical Trial. Circulation. 2019 Nov 26;140(22):1779-1788. doi: 10.1161/CIRCULATIONAHA.119.042622. Epub 2019 Oct 21. PMID 31630538
- [Background] Mol D, Boersma AM, Berger WR, Khan M, de Ruiter GS, Kimman GP, de Groot JR, de Jong JSSG. Intermediate-term outcome of cryoballoon ablation of persistent atrial fibrillation and improvements in quality of life of patients. PLoS One. 2022 Jan 21;17(1):e0261841. doi: 10.1371/journal.pone.0261841. eCollection 2022. PMID 35061716
- [Background] Verma A, Jiang CY, Betts TR, Chen J, Deisenhofer I, Mantovan R, Macle L, Morillo CA, Haverkamp W, Weerasooriya R, Albenque JP, Nardi S, Menardi E, Novak P, Sanders P; STAR AF II Investigators. Approaches to catheter ablation for persistent atrial fibrillation. N Engl J Med. 2015 May 7;372(19):1812-22. doi: 10.1056/NEJMoa1408288. PMID 25946280
- [Background] Tondo C, Iacopino S, Pieragnoli P, Molon G, Verlato R, Curnis A, Landolina M, Allocca G, Arena G, Fassini G, Sciarra L, Luzi M, Manfrin M, Padeletti L; ClinicalService 1STOP Project Investigators. Pulmonary vein isolation cryoablation for patients with persistent and long-standing persistent atrial fibrillation: Clinical outcomes from the real-world multicenter observational project. Heart Rhythm. 2018 Mar;15(3):363-368. doi: 10.1016/j.hrthm.2017.10.038. Epub 2017 Oct 26. PMID 29107190
- [Background] Mansour M, Holmvang G, Sosnovik D, Migrino R, Abbara S, Ruskin J, Keane D. Assessment of pulmonary vein anatomic variability by magnetic resonance imaging: implications for catheter ablation techniques for atrial fibrillation. J Cardiovasc Electrophysiol. 2004 Apr;15(4):387-93. doi: 10.1046/j.1540-8167.2004.03515.x. PMID 15089984
- [Background] Ronsoni RM, Silvestrini TL, Saffi MAL, Leiria TLL. Impact of the left common ostium following pulmonary vein isolation in AF: Systematic review and meta-analysis. J Arrhythm. 2022 Apr 5;38(3):287-298. doi: 10.1002/joa3.12710. eCollection 2022 Jun. PMID 35785389
- [Background] Proietti R, Santangeli P, Di Biase L, Joza J, Bernier ML, Wang Y, Sagone A, Viecca M, Essebag V, Natale A. Comparative effectiveness of wide antral versus ostial pulmonary vein isolation: a systematic review and meta-analysis. Circ Arrhythm Electrophysiol. 2014 Feb;7(1):39-45. doi: 10.1161/CIRCEP.113.000922. Epub 2014 Jan 2. PMID 24385448
- [Background] Reddy VY, Dukkipati SR, Neuzil P, Anic A, Petru J, Funasako M, Cochet H, Minami K, Breskovic T, Sikiric I, Sediva L, Chovanec M, Koruth J, Jais P. Pulsed Field Ablation of Paroxysmal Atrial Fibrillation: 1-Year Outcomes of IMPULSE, PEFCAT, and PEFCAT II. JACC Clin Electrophysiol. 2021 May;7(5):614-627. doi: 10.1016/j.jacep.2021.02.014. Epub 2021 Apr 28. PMID 33933412
- [Background] Sorensen SK, Johannessen A, Worck R, Hansen ML, Hansen J. Radiofrequency Versus Cryoballoon Catheter Ablation for Paroxysmal Atrial Fibrillation: Durability of Pulmonary Vein Isolation and Effect on Atrial Fibrillation Burden: The RACE-AF Randomized Controlled Trial. Circ Arrhythm Electrophysiol. 2021 May;14(5):e009573. doi: 10.1161/CIRCEP.120.009573. Epub 2021 Apr 9. PMID 33835823